CLINICAL TRIAL: NCT01595529
Title: Targeted Clinical Trials to Reduce the Risk of Antimicrobial Resistance The SCOUT Study: "Short Course Therapy for Urinary Tract Infections in Children"
Brief Title: The SCOUT Study: "Short Course Therapy for Urinary Tract Infections in Children"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-0103
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2013-10-22

CONDITIONS: Urinary Tract Infection
Keywords: antibiotic therapy; antimicrobial resistance; children; E.coli; K.pneumoniae; parent study; SCOUT Study; spectrum stool bacteria; stool culture; urinary tract infections
MeSH Terms: conditions — Urinary Tract Infections; Escherichia coli Infections | interventions — Cefixime; Cephalexin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment (Experimental): 5 days of active therapy to match the physician-initiated therapy, Trimethoprim sulfamethoxazole, Cefixime or Cefdinir or Cephalexin (subjects originally receiving Cefdinir will receive Cefixime)
  Interventions: Drug: Cefixime; Drug: Cephalexin; Drug: Trimethoprim/Sulfamethoxazole
- Placebo treatment (Placebo Comparator): 5 days of placebo treatment to match physician-initiated therapy
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cefixime — Cefixime 8 mg/kg/day orally, in 1 dose, with a maximum of 400 mg. Subjects originally receiving Cefdinir will receive Cefixime.
  Arms: Active treatment
Drug: Cephalexin — Cephalexin 50mg/kg/day in 3 divided doses
  Arms: Active treatment
Other: Placebo — Placebo to match the other four active treatments
  Arms: Placebo treatment
Drug: Trimethoprim/Sulfamethoxazole — 8 mg/kg/day of Trimethoprim-sulfamethoxazole (TMP-SMX) orally in 2 divided doses, with a maximum dose of 160 mg twice a day.
  Arms: Active treatment

SUMMARY:
The SCOUT study is a multi-center, centrally randomized, double-blind, placebo-controlled non-inferiority clinical trial. 746 participants will be enrolled over a 4.5 year period. 672 will be evaluated for the study's primary outcome measure. After the first 5 days of primary care physician initiated antimicrobial therapy, patients who are afebrile and asymptomatic will then be randomized (1:1) to the standard course therapy arm of 5 more days of the same antibiotic therapy or the short course therapy arm of a placebo for 5 more days (for 10 days total). The primary objective of this study is to determine if halting antimicrobial therapy in subjects who have exhibited clinical improvement 5 days after starting antibiotic therapy (short course therapy) have the same failure rate (symptomatic UTI) through visit Day 11-14 as subjects who continue to take antibiotics for an additional 5 days (standard course therapy).

DETAILED DESCRIPTION:
The SCOUT Study is a multi-center, centrally randomized, double-blind, placebo-controlled non-inferiority clinical trial of 746 children ages two months (at least 36 weeks gestation from birth for subjects < two years of age) to 10 years with a confirmed diagnosis of a urinary tract infection (UTI) to evaluate 672 for the study's primary outcome measure. UTI is one of the most common serious bacterial infections during childhood. Escherichia coli (E. coli) isolates account for 80-90 percent of all outpatient UTIs in children. Although antibiotics are the first treatment choice for urinary tract infections, antibiotic-resistant strains of E. coli, the most common cause of UTIs, are increasing worldwide. The study will enroll 746 children who have demonstrated clinical improvement five days after starting the originally prescribed antibiotic (afebrile and asymptomatic) and they will be randomized either to the standard-course arm or the short-course arm at a 1:1 ratio. Subjects will be enrolled over approximately a four and a half year period. Study duration for each individual subject will be approximately five weeks. The study product will consist of trimethoprim-sulfamethoxazole (TMP-SMX), cefixime, cefdinir, cephalexin and the corresponding placebos. The primary objective of this study is to determine if halting antimicrobial therapy in subjects who have exhibited clinical improvement 5 days after starting antibiotic therapy (short course therapy) have the same failure rate (symptomatic UTI) through visit Day 11-14 as subjects who continue to take antibiotics for an additional 5 days (standard course therapy). The secondary objectives are: 1) to determine if short-course therapy compared to standard course therapy results in similar numbers of children experiencing a recurrent urinary tract infection (relapse and reinfection; 2) to determine if short-course therapy compared to standard course therapy results in similar numbers of children with asymptomatic bacteriuria; 3) to determine if short-course therapy compared to standard course therapy results in similar numbers of children with gastrointestinal colonization of antimicrobial resistant Escherichia coli (E. coli) and Klebsiella pneumonia (K. pneumoniae); 4) to determine if short-course therapy compared to standard course therapy results in similar numbers of subjects presenting with clinical symptoms that may be related to UTI; 5) to determine if the number of subjects with positive urine culture prior to or at visit Day 11-14 is similar after short-course therapy compared to standard course therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age at randomization: at least two months (at least 36 weeks gestational age for subjects less than two years of age) to 10 years of age (120 months).
2. Confirmed UTI (Urinary Tract Infection) diagnosis.
3. Documented Clinical Improvement at Randomization.

   1. Afebrile: No documented temperature > / = 100.4 degrees Fahrenheit or 38 degrees Celsius (measured anywhere on the body) 24 hours prior to the enrollment visit
   2. Asymptomatic: report NONE of the following symptoms:

      * Symptoms for all children (ages two months to 10 years):

        * Fever (a documented temperature of at least 100.4 degrees Fahrenheit OR 38 degrees Celsius measured anywhere on the body)

          * dysuria
      * Additional symptoms for children > 2 years of age:

        * suprapubic, abdominal, or flank pain or tenderness OR
        * urinary urgency, frequency, or hesitancy (defined as an increase in these symptoms from pre-diagnosis conditions)
      * Additional symptoms for children > / = 2 months to 2 years of age:

        * poor feeding OR
        * vomiting
4. Only children who have been prescribed one of the four antibiotics for which a placebo is available will be eligible to participate.

   * TMP-SMX; Cefixime; Cefdinir or Cephalexin. (Note a child that received a one-time dose of I.M. or I.V. medication (i.e. in ER or clinic) prior to starting on the one of the four oral medications is eligible for enrollment)
5. Parental or guardian permission (informed consent) and if appropriate, child assent (if > / = seven years of age).

Exclusion Criteria:

1. A urine culture proven infection with a second uropathogen > 10,000 CFU/mL collected via suprapubic aspiration or catheter or > 50,000 CFU/mL collected via clean void.
2. A child hospitalized with a UTI that has the following: concomitant bacteremia associated with the UTI, urosepsis, or is in intensive care.
3. A child whose urine culture reveals an organism that is resistant to the initially prescribed antibiotic.
4. A child with a catheter-associated UTI.
5. A child with known anaphylactic allergies to the study products.
6. A child with phenylketonuria (PKU).
7. A child diagnosed with congenital anomalies of the genitourinary tract.
8. UTI in children with known anatomic abnormalities of the genitourinary tract other than VUR (Vesicoureteral reflux), duplicated collection systems, and hydronephrosis.
9. A child that is not able to take oral medications.
10. Previous surgery of the genitourinary tract (except circumcision in male children).
11. Presence of an immunocompromising condition (e.g., HIV, malignancy, solid-organ transplant recipients, use of chronic corticosteroids or other immunosuppressive agents).
12. Unlikely to complete follow-up (e.g. not available for the two follow-up study visits and the follow-up phone call).
13. A child with a known history of type I hypersensitivity of the study antibiotics to be prescribed .
14. Enrollment in another antibiotic study less than 30 days prior to enrollment visit.
15. Previous enrollment of individuals in this study.
16. Planned enrollment during this study coincides with enrollment in another therapeutic drug study (excluding vaccine).
17. A child with a history of UTI within the past 30 days.
18. A child with known Grade III-V VUR.
19. A child taking antibiotic prophylaxis for any reason.
20. A child who has started Day 6 of the originally prescribed antibiotic treatment.

Ages: 2 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 717 (Actual)
Dates: Start 2012-05-18 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Pittsburgh of UPMC - General Academic Pediatric, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Zaoutis T, Shaikh N, Fisher BT, Coffin SE, Bhatnagar S, Downes KJ, Gerber JS, Shope TR, Martin JM, Muniz GB, Green M, Nagg JP, Myers SR, Mistry RD, O'Connor S, Faig W, Black S, Rowley E, Liston K, Hoberman A. Short-Course Therapy for Urinary Tract Infections in Children: The SCOUT Randomized Clinical Trial. JAMA Pediatr. 2023 Aug 1;177(8):782-789. doi: 10.1001/jamapediatrics.2023.1979. PMID 37358858

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 717 enrolled, 23 did not meet the screening criteria and 1 withdrew consent prior to randomization. 693 subjects were randomized.
Groups:
- Standard Course Treatment: 5 days of active therapy to match the physician-initiated therapy, Trimethoprim sulfamethoxazole, Cefixime or Cefdinir or Cephalexin (subjects originally receiving Cefdinir will receive Cefixime)
  Cefixime: Cefixime 8 mg/kg/day orally, in 1 dose, with a maximum of 400 mg. Subjects originally receiving Cefdinir will receive Cefixime.
  Cephalexin: Cephalexin 50mg/kg/day in 3 divided doses
  Trimethoprim/Sulfamethoxazole: 8 mg/kg/day of Trimethoprim-sulfamethoxazole (TMP-SMX) orally in 2 divided doses, with a maximum dose of 160 mg twice a day.
- Short Course Treatment: 5 days of placebo treatment to match physician-initiated therapy
  Placebo: Placebo to match the other four active treatments
Period: Overall Study
Arm/Group | Standard Course Treatment | Short Course Treatment
Started (Randomized.) | 348 | 345
Treated | 337 | 340
Evaluated for Primary Endpoint, ITT (Participants taking at least one dose of treatment from Day 6-10, evaluated at or failed before TOC.) | 328 | 336
ITT Without Treatment Failure (This group was used to evaluate recurrent infection.) | 326 | 322
ITT With Stool Sample at TOC (This group was used to evaluate colonization with antibiotic-resistant E. coli and K. pneumoniae.) | 298 | 310
Per-protocol, Completed 80% of Dose (Participants who completed more than 80% of the prescribed dose between Day 6 and Day 10.) | 308 | 314
Per-protocol Without Treatment Failure (This group was used to evaluate recurrent infection.) | 306 | 305
Per-protocol With Stool Sample at TOC (This group was used to evaluate colonization with antibiotic-resistant E. coli and K. pneumoniae.) | 280 | 289
Completed All Milestones | 318 | 318
Completed (A subject could have completed the study without completing all appointments.) | 324 | 325
Not Completed | 24 | 20
Not completed — Adverse Event | 2 | 0
Not completed — Subject Non-Compliant | 2 | 0
Not completed — Lost to Follow-up | 8 | 14
Not completed — Protocol Violation | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Consent Withdrawn/Voluntary Withdrawal | 3 | 3
Not completed — Administrative Decision | 1 | 0
Not completed — Entry Failure/Screening Failure | 6 | 1

BASELINE CHARACTERISTICS:
Population: Of the 677 treated patients, only 664 were able to be evaluated for the primary endpoint.
  Subject noncompliant: 4 Consent withdrawn: 3 Admin/Inv decision: 2 AE concomitant infection: 2 Lost to follow-up: 1 Protocol violation/deviation: 1
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Course Treatment | Short Course Treatment | Total
Number analyzed (Participants) | 328 | 336 | 664
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.31 (2.71) | 4.16 (2.62) | 4.23 (2.66)
Age, Customized [Count of Participants; unit: Participants]
  Age: 2 months - 35 months | 95 | 89 | 184
  Age: 3 - 6 years | 148 | 177 | 325
  Age: 7 - 10 years | 85 | 70 | 155
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 316 | 323 | 639
  Male | 12 | 13 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 217 | 210 | 427
  Race: Black/African American | 73 | 83 | 156
  Race: Asian | 5 | 8 | 13
  Race: Native Hawaiian/Other Pacific Islander | 0 | 2 | 2
  Race: American Indian/Alaska Native | 0 | 2 | 2
  Race: Multi-Racial | 23 | 25 | 48
  Race: Other | 9 | 6 | 15
  Race: Unknown | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 33 | 27 | 60
  Ethnicity: Not Hispanic | 295 | 309 | 604

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Efficacy Based on Symptomatic Urinary Tract Infection (UTI) Between Short-course and Standard-course of Antibiotics.
Description: A subject will be categorized as a treatment failure, if he/she has a symptomatic UTI in period between Day 6 through the Day 11 - 14 Test of Cure (TOC) Visit:
  1. Symptoms
     * Symptoms for all subjects (ages two months to 10 years): fever (a documented temperature of at least 100.4 °F OR 38°C measured anywhere on the body) ,dysuria
     * Additional symptoms for subjects > 2 years of age: suprapubic, abdominal, or flank pain or tenderness OR urinary urgency, frequency, or hesitancy (defined as an increase in these symptoms from pre-diagnosis conditions)
     * Additional symptoms for subjects = 2 months to 2 years of age: poor feeding OR vomiting AND
  2. Pyuria on urinalysis AND
  3. Culture proven infection with a single uropathogen NOTE: As per the above criteria, asymptomatic subjects (including subjects assessed as having asymptomatic bacteriuria) at the Day 11-14 TOC visit will NOT be considered a treatment failure for the primary outcome measure.
Time Frame: Day 11 through Day 14
Population: Intent to treat population, ITT. All subjects taking at least one dose of study treatment between Day 6 and Day 10 who have been evaluated for treatment success at TOC or have failed prior to TOC.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Course Treatment | Short Course Treatment
Number analyzed (Participants) | 328 | 336
Participants | 2 | 14
Statistical Analysis 1: Comparison: Standard Course Treatment vs Short Course Treatment; Test type: Non-Inferiority — The primary analysis was a non-inferiority test comparing the proportion of subjects with symptomatic UTIs at the TOC visit to evaluate whether the difference was within the 5% equivalence interval. This test was conducted by calculating the one-sided 95% upper confidence limit for the difference in symptomatic UTI (treatment failure) rate. If this limit was less than or equal to the equivalence interval (0.05), then would conclude that short course therapy is not inferior to standard therapy; Risk Difference (RD) = 0.035569, 95% CI 1-sided [upper limit 0.054844]

2. Primary Outcome: Comparison of Efficacy Based on Symptomatic Urinary Tract Infection (UTI) Between Short-course and Standard-course of Antibiotics. Per-protocol Population.
Description: as for outcome 1
Time Frame: Day 11 through Day 14
Population: Per-protocol Population (PP): The enrolled subjects who were adherent to their assigned study regimen and completed more than 80% of the prescribed dose between Day 6 and Day 10 (per-protocol population).
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Course Treatment | Short Course Treatment
Number analyzed (Participants) | 308 | 314
Participants | 2 | 9
Statistical Analysis 1: Comparison: Standard Course Treatment vs Short Course Treatment; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.022169, 95% CI 1-sided [upper limit 0.03939]

3. Secondary Outcome: Comparison of Number of Subjects That Have a Recurrent Infection (Includes a Relapse UTI or a Reinfection) Following Short-course Versus Standard-course of Antibiotics.
Time Frame: Day 11 through Day 44
Population: Subjects in the ITT population who did not experience a treatment failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Course Treatment | Short Course Treatment
Number analyzed (Participants) | 326 | 322
Participants | 12 | 13
Statistical Analysis 1: Comparison: Standard Course Treatment vs Short Course Treatment; Test type: Superiority; Risk Difference (RD) = -0.00356, 95% CI 2-sided [-0.03323 to 0.026102]

4. Secondary Outcome: Comparison of Number of Subjects That Have a Recurrent Infection (Includes a Relapse UTI or a Reinfection) Following Short-course Versus Standard-course of Antibiotics. Per-protocol Population.
Time Frame: Day 11 through Day 44
Population: Subjects in the per-protocol population who did not experience a treatment failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Course Treatment | Short Course Treatment
Number analyzed (Participants) | 306 | 305
Participants | 10 | 13
Statistical Analysis 1: Comparison: Standard Course Treatment vs Short Course Treatment; Test type: Superiority; Risk Difference (RD) = -0.00994, 95% CI 2-sided [-0.04012 to 0.020236]

5. Secondary Outcome: Comparison of the Number of Subjects That Become Colonized With Antimicrobial Resistant Escherichia Coli (E. Coli) and Klebsiella Pneumoniae (K. Pneumoniae) in the Gastrointestinal Tract Following Short-course Versus Standard Course of Antibiotics.
Description: A child would have emergent antibiotic resistance if they:
  1. Had no antibiotic-resistant E.coli or K.pneumoniae at enrollment but one or both are now present. OR
  2. Had either antibiotic-resistant E.coli or K.pneumoniae at enrollment but now the other antibiotic-resistant organism is present OR
  3. Had antibiotic-resistant E.coli and/or K.pneumoniae at enrollment, but have now developed resistance to new antibiotics in either organism.
Time Frame: Day 11 through Day 30
Population: Subjects in the ITT population who have a stool sample at TOC visit. Some treatment failures will not have a sample collected at TOC because they failed prior to TOC. Treatment failures without the sample at TOC are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Course Treatment | Short Course Treatment
Number analyzed (Participants) | 298 | 310
Participants
  Test of Cure Visit (Day 11-14) | 22 | 31
  Outcome Assessment Visit (Day 24-30) | 23 | 28
Statistical Analysis 1: Comparison: Standard Course Treatment vs Short Course Treatment; At Test of Cure Visit; Test type: Superiority; p = 0.2282, Chi-squared
Statistical Analysis 2: Comparison: Standard Course Treatment vs Short Course Treatment; At Outcome Assessment Visit; Test type: Superiority; p = 0.4876, Chi-squared

6. Secondary Outcome: Comparison of the Number of Subjects That Become Colonized With Antimicrobial Resistant E. Coli and K. Pneumoniae in the Gastrointestinal Tract Following Short-course Versus Standard Course of Antibiotics. Per-protocol Population.
Description: as for outcome 5
Time Frame: Day 11 through Day 30
Population: Subjects in the ITT population who have a stool sample at TOC visit. Some treatment failures will not have a sample collected at TOC because they failed prior to TOC. Treatment failures without the sample at TOC would be excluded from the Antibiotic Resistant ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Course Treatment | Short Course Treatment
Number analyzed (Participants) | 280 | 289
Participants
  Test of Cure Visit (Day 11-14) | 22 | 28
  Outcome Assessment Visit (Day 24-30) | 23 | 23
Statistical Analysis 1: Comparison: Standard Course Treatment vs Short Course Treatment; At Test of Cure Visit; Test type: Superiority; p = 0.4184, Chi-squared
Statistical Analysis 2: Comparison: Standard Course Treatment vs Short Course Treatment; At Outcome Assessment Visit; Test type: Superiority; p = 0.9782, Chi-squared

7. Secondary Outcome: Comparison of the Number of Subjects With Asymptomatic Bacteriuria Following Short-course Versus Standard-course of Antibiotics.
Description: Asymptomatic Bacteriuria is defined in any SCOUT subject by:
  1. Absence of symptoms attributable to UTI including fever AND/OR the following:
     * Symptoms for all children (ages two months to 10 years):
       * fever (a documented temperature of at least 100.4 °F OR 38°C measured anywhere on the body)
       * dysuria
     * Additional symptoms for children > 2 years of age:
       * suprapubic, abdominal, or flank pain or tenderness OR
       * urinary urgency, frequency, or hesitancy (defined as an increase in these symptoms from pre-diagnosis conditions)
     * Additional symptoms for children = 2 months to 2 years of age:
       * poor feeding OR
       * vomiting AND
  2. A positive urine culture
     * 5 x 104 CFU/mL (catheterized or suprapubic aspiration urine specimen) OR
     * >105 CFU/mL (clean void specimen).
Time Frame: Day 11 through Day 14
Population: Intent-to-treat (ITT) Population: All subjects taking at least one dose of study treatment between Day 6 and Day 10 who have been evaluated for treatment success at TOC or have failed prior to TOC.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Course Treatment | Short Course Treatment
Number analyzed (Participants) | 328 | 336
Participants | 11 | 29
Statistical Analysis 1: Comparison: Standard Course Treatment vs Short Course Treatment; Test type: Superiority; Risk Difference (RD) = -0.05277, 95% CI 2-sided [-0.08857 to -0.01698]

8. Secondary Outcome: Comparison of the Number of Subjects With Asymptomatic Bacteriuria Following Short-course Versus Standard-course of Antibiotics. Per-protocol Population.
Description: as for outcome 7
Time Frame: Day 11 through Day 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Course Treatment | Short Course Treatment
Number analyzed (Participants) | 308 | 314
Participants | 11 | 29
Statistical Analysis 1: Comparison: Standard Course Treatment vs Short Course Treatment; Test type: Superiority; Risk Difference (RD) = -0.05664, 95% CI 2-sided [-0.09479 to -0.01850]

9. Secondary Outcome: Comparison of the Number of Subjects With Clinical Symptoms That May be Related to a UTI Following Short-course Versus Standard-course of Antibiotics.
Time Frame: Up to Day 14
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Course Treatment | Short Course Treatment
Number analyzed (Participants) | 328 | 336
Participants | 30 | 41
Statistical Analysis 1: Comparison: Standard Course Treatment vs Short Course Treatment; Test type: Superiority; Risk Difference (RD) = -0.03056, 95% CI 2-sided [-0.07744 to 0.016323]

10. Secondary Outcome: Comparison of the Number of Subjects With Clinical Symptoms That May be Related to a UTI Following Short-course Versus Standard-course of Antibiotics. Per-protocol Population
Time Frame: Up to Day 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Course Treatment | Short Course Treatment
Number analyzed (Participants) | 308 | 314
Participants | 29 | 33
Statistical Analysis 1: Comparison: Standard Course Treatment vs Short Course Treatment; Test type: Superiority; Risk Difference (RD) = -0.01094, 95% CI 2-sided [-0.0580 to 0.036117]

11. Secondary Outcome: Comparison of the Number of Subjects With Positive Urine Cultures Following Short-course Versus Standard-course of Antibiotics.
Time Frame: Up to Day 14
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Course Treatment | Short Course Treatment
Number analyzed (Participants) | 328 | 336
Participants | 6 | 41
Statistical Analysis 1: Comparison: Standard Course Treatment vs Short Course Treatment; Test type: Superiority; Risk Difference (RD) = -0.10373, 95% CI 2-sided [-0.14161 to -0.06585]

12. Secondary Outcome: Comparison of the Number of Subjects With Positive Urine Cultures Following Short-course Versus Standard-course of Antibiotics. Per-protocol Population.
Time Frame: Up to Day 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Course Treatment | Short Course Treatment
Number analyzed (Participants) | 308 | 314
Participants | 6 | 35
Statistical Analysis 1: Comparison: Standard Course Treatment vs Short Course Treatment; Test type: Superiority; Risk Difference (RD) = -0.09198, 95% CI 2-sided [-0.13006 to -0.05391]

ADVERSE EVENTS:
Time Frame: Day 6 to Day 44 Follow-up Phone Call
Arm/Group | Standard Course Treatment | Short Course Treatment
All-Cause Mortality (participants affected / at risk) | 0/328 | 0/336
Serious Adverse Events (participants affected / at risk) | 2/328 | 4/336
Other Adverse Events (participants affected / at risk) | 155/328 | 147/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Course Treatment (N=328) | Short Course Treatment (N=336)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
URETHRAL VALVES (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Course Treatment (N=328) | Short Course Treatment (N=336)
DIARRHOEA (Gastrointestinal disorders) | 42 | 34
PYREXIA (General disorders) | 15 | 18
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 12 | 16
VOMITING (Gastrointestinal disorders) | 11 | 20
COUGH (Respiratory, thoracic and mediastinal disorders) | 21 | 23
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 10 | 12
RASH (Skin and subcutaneous tissue disorders) | 11 | 12
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 | 10
CONSTIPATION (Gastrointestinal disorders) | 8 | 7
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 7 | 5
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 4 | 4
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 4
VIRAL INFECTION (Infections and infestations) | 1 | 4
GASTROENERITIS (Infections and infestations) | 4 | 0
NASOPHARYNGITIS (Infections and infestations) | 2 | 5
OTITIS MEDIA ACUTE (Infections and infestations) | 5 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 5
TEETHING (Gastrointestinal disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT01595529/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT01595529/SAP_001.pdf